CLINICAL TRIAL: NCT02882984
Title: Comparing Whole Brain Radiation With Hypofractionated Stereotactic RadioSurgery (HFSRS) in Patients With NSCL Brain Metastases
Brief Title: Hypofractionated Brain Radiation In EGFR Mutated Adenocarcinoma Cranial Disease (Hybrid)
Acronym: Hybrid
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, ming zeng, MD, Director of Cancer Center, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hybrid
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Stage IV EGFR Mutated NSCL With Brain Metastases
MeSH Terms: interventions — Gefitinib; Erlotinib Hydrochloride; icotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBRT along with TKI (Active Comparator): Drug: EGFR-TKI
  Gefitinib 250mg po qd or Tarceva 150mg po qd or Icotinib 125mg po tid
  Other Name: Gefitinib/Tarceva/Icotinib
  Radiation: whole brain radiotherapy
  3750Gy/15F
  Other Name: WBRT
  Interventions: Drug: Gefitinib 250mg po qd or Tarceva 150mg po qd or Icotinib 125mg po tid Other Name: Gefitinib/Tarceva/Icotinib; Radiation: WBRT
- HFSRS with EGFR TKI (Experimental): Drug: EGFR-TKI
  Gefitinib 250mg po qd or Tarceva 150mg po qd or Icotinib 125mg po tid
  Other Name: Gefitinib/Tarceva/Icotinib
  Radiation: whole brain radiotherapy
  25 to 40 Gy/5F
  Other Name: HFSRS
  Interventions: Drug: Gefitinib 250mg po qd or Tarceva 150mg po qd or Icotinib 125mg po tid Other Name: Gefitinib/Tarceva/Icotinib; Radiation: HFSRS

INTERVENTIONS:
Drug: Gefitinib 250mg po qd or Tarceva 150mg po qd or Icotinib 125mg po tid Other Name: Gefitinib/Tarceva/Icotinib — radiation given along with one of kind TKI
  Other Names: EGFR-TKI
Radiation: WBRT — 3750 cGy in 15 fractions given within 3 weeks time.
  Arms: WBRT along with TKI
Radiation: HFSRS — All HFSRS given in 5 fractions. dose per fraction ranges from 5 to 8 Gy depending on the target volume and organs at risk tolerance.
  Arms: HFSRS with EGFR TKI

SUMMARY:
A multi-center phase III randomized controlled study to evaluate the efficacy of Hypofractionated SRS (HFSRS) along with EGFR-TKI in patients with brain metastasis from non-small cell lung cancer (NSCLC). Assuming that HFSRS is not inferior to EGFR-TKI concurrent with whole brain radiotherapy (WBRT), the primary end point is intracranial PFS (iPFS), while secondary outcomes included overall survival (OS), evaluation of cognitive function, quality of life (QoL) and adverse events.

DETAILED DESCRIPTION:
WBRT remains to be standard of care for NSCL patients. Long term survival from WBRT may have noticeable cognitive dysfunction. The EGFR TKI has reasonable control for intracranial disease, but the duration of EGFR TKI control disease is variable due to tendency of drug resistance. To maintain intracranial disease control and improve cognitive function, the investigators propose using hypofractionated SRS in multiple brain metastases or large brain lesions alone with TKI.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small cell lung cancer (NSCLC);
* Diagnosis of brain metastases on a Gadolinium-enhanced MRI.
* More than 3 sites of intracranial metastases, or the longest diameter of the intracranial lesion is more than 4 cm.
* Positive EGFR mutation.
* Life expectancy ≥3months.
* Have one or more measurable encephalic lesions according to RECIST.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L.
* Adequate renal function: Serum creatinine ≤1.5 x ULN, or ≥ 50 ml/min.
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) and Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.
* Female subjects should not be pregnant.
* All human subjects should able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Written informed consent provided.

Exclusion Criteria:

* Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.
* CSF or MRI findings consistent with metastases of spinal cord, meninges or meningeal.
* Allergic to Icotinib.
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
* Pregnancy or breast-feeding women.
* Participate in the other anti-tumor clinical trials in 4 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
iPFS | 18 months
  intracranial progression-free survival

SECONDARY OUTCOMES:
cognitive function | 18 month
  Neurocognitive effects evaluated according to Mini-Mental Status Examination Evaluated according to Mini-Mental Status Examination
Overall survival (OS) | 18 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zeng, MD PhD, Study Chair — Sichuan Provincial People Hospital, Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan PPH, Cancer Center, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided